CLINICAL TRIAL: NCT02044185
Title: Observational Study for Clinical Implications of HMGB1 (High-mobility Group Protein B1) in Patients Treated With Chemotherapy or Hematopoietic Stem Cell Transplantation
Brief Title: Clinical Implications of HMGB1 in Patients Treated With Chemotherapy or Hematopoietic Stem Cell Transplantation
Acronym: CHIP-SCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, JEON YOUNG-WOO, medical doctor, fellowship, Seoul St. Mary's Hospital
Other Study IDs: CMC-SGC-Lymphoma-LAB-01
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Acute Graft-versus-host Disease
Keywords: HMGB1 Protein; Graft versus Host Disease; Immunosuppressive Agents; oral mucositis
MeSH Terms: conditions — Graft vs Host Disease; Stomatitis | interventions — Whole-Body Irradiation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma biopsy tissue samples of colon
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high dose chemotherapy: group of using myeloablation regimen, autologous stell cell transplantation
  Interventions: Drug: salvage chemotherapy, total body irradiation
- control group: normal population with health screening
  Interventions: Drug: salvage chemotherapy, total body irradiation

INTERVENTIONS:
Drug: salvage chemotherapy, total body irradiation — there are no direct interventions to our patients.

SUMMARY:
Acute Graft-versus-host disease(aGVDH) after allogeneic hematopoietic stem cell transplantation is one of the meaningful issues in aspect of patient's recovery and survival. in recent years, the understanding of the pathology of GVHD is much important to prevent or treat aGVHD. additionally, (oral) mucositis is one of the problems in patients with high dose chemotherapy, and mucositis by high-dose chemotherapy is related to HMGB-1 as proinflamtory cytokines. HMGB1 is a nuclear protein acts as a transcription factor, but, if it was released to the outside of cells by damaged cell or necrotic tissues, it works as cytokines for promoter of inflammation and cancers. at this point, there are no reported articles about correlation of HMGB1 and aGVHD in human. recently, we have seen excessive secretion of serum HMGB1 in mouse model, then base on this results, we will check correlation of HMGB1 and aGVHD/ oral mucositis in human.

DETAILED DESCRIPTION:
1. materials 1) inclusion criteria

   1. over 18-year-old
   2. patients with myeloablative conditioning regimen
   3. autologous transplant
   4. patients with confirmation of acute GVHD as over grade II
   5. patients with salvage chemotherapy

      2) exclusion criteria

   <!-- -->

   1. old age ( over 60-year-old)
   2. patients with reduced intensity stem cell transplantation
2. method 1) check the serum level of HMGB1, TNF-a, IL-1b, IL-6, Th1, Th2, Th17, FoxP3 on 7-day before transplant day(D-7), transplant day(D0), 7-day after transplant(D+7), D+14, D+21. 2) check the immunohistochemistry level of tissue in diagnosed aGVHD ( performed sigmoidoscopy and random biopsy of gut is routine process in our center) 3) check the oral mucositis grades (using WHO grading system, NCI -CTC ver.3 scoring system)
3. analysis 1) student t-test , chi-square test 2) survival analysis

ELIGIBILITY:
1. Inclusion Criteria:

   1. over 18-year-old
   2. patients with myeloablative conditioning regimen
   3. autologous transplant
   4. patients with confirmation of acute GVHD as over grade II
   5. patients with salvage chemotherapy
2. Exclusion Criteria:

   1. very old age ( over 75-year-old)
   2. patients with reduced intensity stem cell transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. patients with bone marrow transplantation of patients with acute leukemia, lymphoma in patients group
  2. normal populations in Health Promotion Center in control group
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
comparison of serum HMGB1 level before and after diagnosed acute GVHD | 6 months
  day 7 before stem cell transplantation(SCT), day 0, day 7, 14 after SCT, and date of diagnosed acute GVHD in all patients.

SECONDARY OUTCOMES:
serum level of immunosuppressive drugs in patients with acute GVHD | 3 months
  day 7 before stem cell transplantation(SCT), day 0, day 7, 14 after SCT, and date of diagnosed acute GVHD in all patients.

OTHER OUTCOMES:
tissue IHC stain level of biopsy samples of diagnosed acute GVHD | if patients diagnosed with acute GVHD will be performed random biopy of colon or stomach.
oral mucositis | 1 month
  find-out the correlation HMGB1 level and oral mucositis grading

CONTACTS AND LOCATIONS:
Overall Officials: seok-goo CHO, M.D,Ph.D, Study Chair — The Catholic University of Korea
Locations (1):
- Seoul St.Mary's hospital, Seoul, South Korea

REFERENCES:
- [Background] Brennan TV, Lin L, Huang X, Cardona DM, Li Z, Dredge K, Chao NJ, Yang Y. Heparan sulfate, an endogenous TLR4 agonist, promotes acute GVHD after allogeneic stem cell transplantation. Blood. 2012 Oct 4;120(14):2899-908. doi: 10.1182/blood-2011-07-368720. Epub 2012 Jul 3. PMID 22760779
- [Background] Kornblit B, Masmas T, Petersen SL, Madsen HO, Heilmann C, Schejbel L, Sengelov H, Muller K, Garred P, Vindelov L. Association of HMGB1 polymorphisms with outcome after allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2010 Feb;16(2):239-52. doi: 10.1016/j.bbmt.2009.10.002. Epub 2009 Oct 9. PMID 19819342
- [Background] Jube S, Rivera ZS, Bianchi ME, Powers A, Wang E, Pagano I, Pass HI, Gaudino G, Carbone M, Yang H. Cancer cell secretion of the DAMP protein HMGB1 supports progression in malignant mesothelioma. Cancer Res. 2012 Jul 1;72(13):3290-301. doi: 10.1158/0008-5472.CAN-11-3481. Epub 2012 May 2. PMID 22552293
- [Background] Kang R, Zhang Q, Zeh HJ 3rd, Lotze MT, Tang D. HMGB1 in cancer: good, bad, or both? Clin Cancer Res. 2013 Aug 1;19(15):4046-57. doi: 10.1158/1078-0432.CCR-13-0495. Epub 2013 May 30. PMID 23723299